CLINICAL TRIAL: NCT03542890
Title: Comparison Between Baska and I-gel in Controlled Mechanically Ventilated Females Undergoing Vaginal Surgeries
Brief Title: Respiration and The Airway With Laryngeal Masks
Status: Completed | Type: Observational
Sponsor: Reham Ali Abdelhaleem Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Reham Ali Abdelhaleem Abdelrahman, Anesthesia Lecturer, Cairo University
Organization: Cairo University (Other)
Other Study IDs: BM2008
Record Dates: First submitted 2018-04-17; First posted 2018-05-31 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Supraglottic Airway Devices
Keywords: Anesthesia, General; Baska; I-gel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Baska Mask: It has a non-inflatable cuff, which is moulded to take up the shape of the supraglottic airway, potentially reducing the risk of oropharyngeal tissue and/or nerve damage induced by cuff over inflation, a known complication with other supraglottic airways.
  Interventions: Device: Baska Mask
- I-gel: The I-gel is a single use (SADs) composed of a soft ,gel-like, non-inflatable cuff made from a thermoplastic elastomer. It has a widened , flattened stem with a rigid bite block that acts as a buccal stabilizer to reduce axial rotation and mal-positioning and a port for gastric tube insertion. It is a latex free device that does not require digital insertion into mouth of patient.
  Interventions: Device: I-gel

INTERVENTIONS:
Device: Baska Mask — used in adult low risk females undergoing elective gynecological operations
  Groups: Baska Mask
Device: I-gel — used in adult low risk females undergoing elective gynecological operations
  Groups: I-gel

SUMMARY:
Baska® mask (Proact Medical Systems, Frenchs Forest NSW, Australia) is displayed in figure 1 which is the latest addition to an array of supra-glottic airway devices in clinical use. It has a non-inflatable cuff, which is moulded to take up the shape of the supraglottic airway, potentially reducing the risk of oropharyngeal tissue and/or nerve damage induced by cuff over inflation, a known complication with other supraglottic airways. However, the cuff differs from other non-inflatable cuffs in that it is continuous with the central channel of the device. As the pressure increases with positive pressure ventilation ,the cuff itself is inflated which may improve the seal so reducing leak and make ventilation more efficient. The Baska mask has two ports (one for venting and other for gastric tube insertion ), so it incorporates an inlet that fits into the upper oesophagus and the dorsal surface of the cuff is moulded to direct any oropharyngeal contents away from the glottis and towards the side channels to which suction can be attached to facilitate aspiration of this space. These features may reduce the risk of pulmonary aspiration of secretions or gastric contents that accumulate in the supraglottic area. In addition, there is integrated bite-block, which reduces the risk of patients biting and blocking the airway. There is insertion tab which is an extended hand-tab attached to the cuff that permits the operator to control the degree of flexion of the device during the insertion. The Baska® mask is inserted in the neutral head position, which may reduce the need for neck manipulation. Initial experience with Baska®mask has demonstrated it to be a suitable airway device for procedures less than 2 hours or when endotracheal intubation is not required.

I-gel airway (Intersurgical Ltd, Workingham, Berkshire,United Kingdom) is displayed in figure 2 which is second generation supraglottic airway devices (SADs) that was introduced in 2007. The I-gel is a single use (SADs) composed of a soft ,gel-like, non-inflatable cuff made from a thermoplastic elastomer. It has a widened , flattened stem with a rigid bite block that acts as a buccal stabilizer to reduce axial rotation and mal-positioning and a port for gastric tube insertion. It is a latex free device that does not require digital insertion into mouth of patient. With an epiglottic rest and wider and shorter stem, the I-gel gives an optimal view of the glottis with a fiber- optic scope so a shorter tube is ideal for endotracheal tube placement. Moreover, I-gel can be inserted as fast as classic LMA (Laryngeal Mask Airway) with adequate ventilation in patients and has no major airway complications. Therefore, it could be a good alternative to classic LMA in emergency airway management or general anesthesia.

DETAILED DESCRIPTION:
The study will be carried on adult female patients to reduce variability in size of the chosen device to enable the investigators to analyze the performance parameters of the two devices with greater authority. The study will be done on anesthetized paralyzed adult female patients undergoing elective gynecological operations that require neuromuscular block but not necessarily tracheal intubation. The investigators will recruit 60 adult female(18-55 years old, ASAI&II) patients to a prospective randomized crossover clinical trial. Patients with history of upper respiratory tract infections, obstructive sleep apnea , potentially full stomach( trauma, morbid obesity BMI> 35, pregnancy, history of gastric regurgitation and heart burn), those with esophageal reflux (hiatus hernia), and those of coagulation disorders will be excluded from the study. All patients will be assessed pre-operatively El-Ganzouri airway score to assess the expected difficulty of intubation and patients with airway scores ≥ 5 will be excluded from the study.The patients will be randomly allocated into two groups(the Baska Mask group & the I-gel group; each group is 30 patients) using computer generated program . An online randomization program (http://www.randomizer.org) will be used to generate random list and to allocate patients into the study groups. Random allocation numbers will be concealed in opaque closed envelops. The patient and investigator assessing study outcomes will all be blinded to the study groups allocation.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients ASA I&II
* Age: 18- 45 years old
* BMI < 35
* Undergoing elective gynecological operations.

Exclusion Criteria:

* Patients with history of upper respiratory tract infections and obstructive sleep apnea.
* Patients who are potentially full stomach such as trauma, pregnancy, history of gastric regurgitation &heart burn, those with esophageal reflux or hiatus hernia.
* Patients with El-Ganzouri airway score ≥ 5 will.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: adult female patients undergoing elective gynecological operations.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | one year
  The airway sealing pressure was the pressure at which leak starts. This leak pressure was calculated as the plateau airway pressure reached while the patient was apneic, and following confirmation of adequate ventilation, the adjustable pressure limit valve was set at 70 cmH2O, the fresh gas flow was set at 6 l.min-1(liter per minute), and the airway pressure was measured on the breathing system pressure gauge. Leak pressure will be defined as the plateau airway pressure that was achieved

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia, Surgical ICU, and Pain Management, Cairo, Egypt